CLINICAL TRIAL: NCT02446873
Title: Cracking the Egg Potential: Improving Young Child Nutrition in Ecuador
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Universidad San Francisco de Quito (Other); Pan American Health Organization (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201409108
Record Dates: First submitted 2015-02-28; First posted 2015-05-18 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Choline Deficiency; Vitamin B-12 Deficiency; Lipids Deficiency; Amino Acids Deficiency
Keywords: children; Ecuador; rural; poor
MeSH Terms: conditions — Choline Deficiency; Vitamin B 12 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control group
- Treatment (Experimental): Egg supplementation
  Interventions: Other: Egg supplementation

INTERVENTIONS:
Other: Egg supplementation — A weekly supply of eggs will be given to the mother in the egg supplementation group with instructions to give the child one egg per day.
  Arms: Treatment

SUMMARY:
The proposed study will fill an important gap in the literature by examining, through a randomized controlled trial, the effect of egg consumption on biochemical markers of choline, vitamin B-12, lipids, and amino acids in young children in a poor rural area of Ecuador. Children from Cotopaxi Province, Ecuador (n=180) will be randomized into one of two groups: 1) intervention, receiving one egg per day for six months; or 2) control. Baseline and endline data on socio-economic factors, and child diet, morbidities, and anthropometry will be collected. Blood will also be drawn from the children at these time points for nutrient biomarker analyses. Through qualitative research the proposed study will provide insight into the attitudes, beliefs, and use of eggs by mothers and other caregivers during the complementary feeding period. The University of San Francisco in Quito (USFQ) will be the lead field coordinator of the research working in partnership with Washington University in St. Louis, Pan-American Health Organization (PAHO) and University of California, Davis.

DETAILED DESCRIPTION:
OBJECTIVES

Objective 1: Test the efficacy daily egg consumption for six months on the macro- and micronutrient status of young children from an indigenous community in Ecuador.

1a. Measure serum concentration of micronutrient biomarkers: choline; betaine; and vitamin B12.

1. b. Measure serum concentrations of macronutrient biomarkers: lipids (total free and esterified); and amino acids.

   Objective 2: Characterize attitudes, beliefs, and use of eggs during the complementary feeding period.
2. a. Describe existing attitudes, beliefs, and use of eggs in young child diets in Ecuador.

2b. Monitor acceptability and tolerance of daily egg consumption among young children.

2c. Assess willingness of caregivers to prepare and give eggs daily to young children.

BACKGROUND AND SIGNIFICANCE

Globally, 165 million children are affected by stunting arising in part from macro- and micronutrient deficiencies during the complementary feeding period; defined as between 6 and 24 months of age. An estimated 200 million children are not meeting their developmental potential in part because of poor nutrition and, in particular, nutrient intake inadequacies. Eggs provide several of these critical nutrients known to be missing in the diets of young children living in poor countries, yet have been largely underutilized in infant and young child nutrition.

Eggs provide essential fatty acids, proteins, and many critical micronutrients at levels above or comparable to other animal source foods, but are relatively more affordable. Eggs are considered a perfect protein source with an amino acid profile against which other proteins are compared. Eggs are also highly concentrated in choline, an important precursor for acetylcholine in neurotransmitter synthesis, phospholipids needed for cell-membrane signaling, and methyl-group donation in the homocysteine production pathway. The evidence for the adverse consequences of choline deficiencies come largely from animal studies, though some studies have shown an association between choline or its metabolites and negative health and development outcomes in children. Only one study has shown that egg consumption among young children can be improved through counseling.

Eggs contribute to dietary diversity. They are one of three animal source food groups together with flesh foods and dairy products, included in the seven food groups used to assess the indicator of minimum dietary diversity in the WHO Indicators for assessing infant and young child feeding practices. However, they are underused in the diets of young children relative to their potential to improve child nutrition, particularly in many African countries but even in Latin America and the Caribbean. Egg consumption the preceding day among children 6 to 8.9 months of age was only 7.3%, 15.8% and 22.8% in Africa, Asia and Latin America, respectively. Among children 12 to 23.9 months of age, consumption increased to only 13.4% in Africa, 33.0% in Asia and 41.8% in Latin America and the Caribbean.

All evidence to date suggests that eggs are underutilized as complementary foods relative to their potential to improve young child nutrition and, in particular, levels of key macro and micronutrients. Research to test the efficacy of dietary egg intakes to improve child nutrition in developing countries is needed. It is also needed to understand attitudes, beliefs and use of eggs during the complementary feeding period.

Significance. Despite the potential of eggs to improve young child nutrition, to our knowledge there have been no randomized controlled trials to test the efficacy of egg consumption to improve the micronutrient status of young children living in developing countries and very little evidence from egg-related interventions. There is also very limited evidence on the attitudes, beliefs, and use of eggs by mothers and other caregivers during the complementary feeding period. Therefore, the proposed study will fill an important gap in the literature by examining, through a randomized controlled trial, the effect of egg consumption on serum concentration of micronutrient biomarkers: B12; choline; and betaine and macronutrient biomarkers: lipids (total free and esterified); and protein nutrition in young children in a poor rural area of Ecuador. Through qualitative research the proposed study will also shed light on the attitudes, beliefs, and use of eggs by mothers and other caregivers during the complementary feeding period.

EXPERIMENTAL DESIGN & METHODS

University of San Francisco in Quito (USFQ) will coordinate all field activities. A randomized controlled trial with a parallel design will be applied. A total of 180 mother-infants pairs enrolled in this study: 90 in the control group; and 90 in the egg intervention group. Inclusion criteria for all infants include: age 6-8 mo; healthy (no fever, congenital heart condition, or egg allergy); singleton birth; and not severely malnourished [weight-for-length z (WLZ) > -3). There will be 180 mothers or if mother is not available, other caregivers of infants (fathers, grandparents, aunts/uncles, siblings, etc.) enrolled.

Participants (recruitment, screening, and consent process). Mothers/primary caregivers and children will be recruited in Pastocalle Parish in Cotopaxi Province of Ecuador, where formative research was conducted to ensure sufficient numbers of infants in this age category. There will be a rolling admission process over a one-year period to ensure sample size is reached, and potentially we will extend recruitment to adjacent parishes. Participants will be recruited through participatory approaches, with the support of local leaders and the active involvement of community stakeholders. There will be an initial stage before recruitment in which the field team will build rapport with caregivers using standardized techniques. Mothers (or other primary caregivers) will be approached and invited to participate with their children in the study. Study staff will verbally explain the rationale for the study, all study procedures and their risks and benefits, and will invite mothers to participate with their children. Eligibility screening will then occur. Screening questions posed to the mother/primary caregiver will include:

* How old are you?
* What is the child's birthday?
* Is the child healthy, without fever or congenital heart condition, and not severely malnourished?
* Does the child have any reactions to eating to eggs, a rash, hives, difficulty breathing?
* Was the birth of this child a singleton birth; he/she does not have a twin or triplet, etc.

If the primary caregiver reports that the child is malnourished and/or the child has the appearance of thinness or other symptoms such as edema, the weight and length of the child will be measured and the weight-for-length Z score determined from the WHO Growth Standards (2006).

Mothers or primary caregivers of children will be given a written informed consent statement in Spanish to read and sign, indicating their consent and consent on behalf of their child. If the mothers/primary caregiver is less than 18 years of age, informed consent process will be sought from their parents or guardians. Participants with limited literacy will be offered the option to have the statement read to them. Caregivers will be invited to ask any questions about the nature of the study during this time. A potential participant will have approximately one week to decide whether or not to participate and thus, have the opportunity to discuss with family and friends.

Study field procedures. Children will be randomized through a computer-generated number sequence program to one of two comparison groups in a 1:1 ratio: 1) control; and 2) egg supplementation.

The baseline survey will first be administered to all mothers/primary caregivers in community centers, health care posts or nurseries on assigned dates. Household level socioeconomic, demographic, water, hygiene, and sanitation information will be collected. Child dietary intake data will be collected using a food frequency questionnaire of commonly used complementary foods, supplemented with targeted questions about child and household egg consumption patterns. Morbidities will be assessed using a two-week recall, with particular focus on respiratory infections given its high prevalence in this population and any symptoms that might be associated with egg allergies. Anthropometric measures of child length and weight will then be taken using international protocols. Phlebotomists from an experienced and well-equipped laboratory in Ecuador, NETLAB, will collect 3 ml of blood from children. A numbing cream will be used for the children.

A weekly supply of eggs will be given to the mother in the egg supplementation group with instructions to give the child one egg per day. Additional messages will be communicated regarding hygiene practices and egg handling and preparation. Eggs will not require refrigeration, but will need to be stored in a cool location. Mothers/caregivers from the control group will be provided vouchers for 6 months of eggs after the completion of the intervention study. All mothers will receive an attendance card that will track participation in study events including baseline and endline visits and qualitative assessment as appropriate. At the completion of the study, all mothers will receive a small personal care gift (lotion or perfume) in appreciation for their contributions.

Motivational workshops will periodically be held by the study coordinator and team to receive feedback from the participants and continue to provide rationale for study participation. These workshops effectively engage caregivers in the study and can minimize losses-to-follow-up. As well, regular meetings with community leaders and health workers will be held to communicate and dialogue about study progress and findings.

Eggs will be purchased locally in Pastocalle and distributed to families on a weekly basis by the study team. (The Food and Agriculture Organization (FAO) will potentially support USFQ to implement a poultry development project that could linked with this study. With technical support from Ministry of Agriculture extension workers, families from Pastocalle will receive and raise chickens for laying eggs.) Eggs for this study will be purchased from these households and an already established project of egg production developed through the Parish Council to support individuals with disabilities.

The study coordinator and enumerator team will contact mothers/primary caregivers lost to follow-up by mobile phones, visits, and through family members and friends, in order to encourage them to return to the study and to collect information about the reasons they have left the study.

Nutrient biomarkers: Nutrient biomarkers assessed for this study will include vitamin B12, choline, betaine, lipids and amino acids. NETLAB in Quito, Ecuador will be responsible for: 1) collecting the blood samples; 2) processing and completing the extraction process for choline/betaine, lipids and amino acids; 3) shipping these samples to Washington University Biomedical Mass Spectrometry Resource Facility; and 4) completing the assay for vitamin B12. Trained phlebotomists will travel to Pastocalle and surrounding parishes periodically to collect blood samples (3 mL from each child). The ethylenediaminetetraacetic acid (EDTA) plasma will be obtained by collecting blood into Vacutainer Tubes marked with participant ID numbers only. The samples will be placed on ice and transported to the NETLAB facility in Quito.

Samples will be processed and the extraction completed for choline, betaine, lipids, and amino acids. For the choline and betaine analytes, an aliquot of plasma is mixed with acetonitrile containing d9-choline and d9-betaine. The acetonitrile extracts are centrifuged, the supernatant is transferred to a micro-centrifuge tube, and dried to completion under nitrogen gas. The micro-centrifuge tube is labeled with participant ID# and date of collection. An extraction process is also completed for processing the lipids and amino acids. These extracted samples will then be shipped on dry ice to Washington University Biomedical Mass Spectrometry Resource Facility in St. Louis, MO by Globalex shipping company. The choline and betaine assays will be tested using LC/MS/MS protocol (Appendix 1). The remaining sample aliquots will be frozen at -80 degrees C. Vitamin B12 will later be tested using a competitive chemiluminescent enzyme immunoassay solid phase.

Qualitative research. Similar qualitative research techniques will be applied here as were used for Focused Ethnographic Studies (FES). The qualitative method is based on grounded theory. Grounded theory is a unique form of qualitative analysis in that it has an inductive orientation for constructing theory out of a systematic analysis of collected data. In-depth interviews and focus groups will be conducted with mothers, grandmothers, and other caregivers, as well as local health care providers, community leaders, and egg producers to understand attitudes, perceptions and use of eggs for young child nutrition.

Structured observations will be conducted in the homesteads of consenting caregivers and child care centers to examine environmental factors, chicken rearing practices, and complementary food storage and egg preparation and feeding practices. Additionally, we follow a combination of three methods for the analysis of collected qualitative data: coding in three stages; abductive reasoning; and schemes generation. Of these three, the core method is the coding on three stages. First, open coding identifies the basic concepts in individual responses. Second, axial coding is developed through the generation of categories and properties that emerge from the pattern of responses and which produces relations between categories and properties. Third, selective coding integrates and refines the main topics and the interrelations between them. Coding will be done by USFQ, with support from investigators from UCD and PAHO to triangulate for quality control.

Data management. USFQ will be responsible for data management of data collected in Pastocalle and at NETLAB (with UC-Davis), and Washington University will be responsible for data generated at the Biomedical Mass Spectrometry Resource Facility. Data entry will be initiated early and continue throughout the study to minimize errors and increase the likelihood of accurate and comprehensive reporting. When potential errors or missing data are identified, managers will inquire with enumerators and caregivers/mothers to either provide appropriate responses or explanatory notes in the data set. Double data entry will be conducted on a sub-set of surveys to check for entry error.

Sample size and statistical analysis. Sample size was estimated based on hypothesized change (difference-in-difference with control) in plasma vitamin B12 concentration of 59.4 pmol/L over the 6 month period based on other previous findings of vitamin B12 supplementation and the variability in vitamin B12 status among infants. This nutrient was selected for sample size calculation because sufficient data was available to estimate variability and potential effects from egg consumption in contrast to the other nutrients that will be studied. We estimate requiring 90 children per group assuming a 20% attrition rate.

Descriptive statistics will first be applied to examine characteristics of the sample, and the primary and secondary outcomes. Univariate tests, including chi squared and t-tests, will then be applied to compare characteristics across trial arms and examine cross-sectional differences in the outcome variables at baseline and endline. Longitudinal modeling for the primary biomarker outcomes (continuous serum/plasma nutrient concentration markers) and secondary growth (LAZ, WAZ, WLZ) and morbidity outcomes (days with diarrhea) will be conducted using generalized least squares (GLS) with random effects. Logit models will be applied to examine adjusted odds of threshold outcomes (nutrient deficiencies, stunting, underweight, wasting, respiratory infection, etc.). All inference analyses for the efficacy of eggs will use intention-to-treat. Quantitative data analyses were performed with STATA software (version 11.1; StataCorp, College Station, TX).

For qualitative data analyses, interview transcripts will be uploaded into Nvivo10 software and coded for themes. Top-line themes will be sub-divided into more detailed categories according to participants' responses in the interviews. Analyses of these categories and themes reveal patterns in the interview data that form the basis of the qualitative findings. A framework matrix analysis of a subset of interviews in the two study arms analyzing key themes will be applied to investigate any systematic differences in responses across study arms.

To measure micronutrient intakes against normative levels of adequacy, the full probability approach will be used. This method allows for a more comprehensive estimate of inadequacy risk across the entire distribution of intakes when compared to a simple cut-point approach in which intakes above and below a threshold level are estimated. Child micronutrient intake will be standardized by subtracting the estimated average requirement (EAR) of the reference distribution and then dividing by the SD of the reference distribution. The resulting number will be compared to a standard normal distribution to obtain the probability of inadequacy, the area to the right under the standard normal curve, and averaged across the sample.

Profile of the Target Population. The target population for this study will be infants ages 6-8 months old from the Pastocalle Parish, which is populated mainly by indigenous communities, in Cotopaxi Province of Ecuador. Findings from a national health and nutrition survey, Encuesta Natcional de Salud y Nutriciόn (ENSANUT-ECU) showed 25.3% of children ages 0-5 years nationally, and 42.3% of indigenous children were stunted (HAZ<-2). Other indicators from this study further demonstrated the nutritional vulnerabilities of indigenous, young children in Ecuador. Prevalences of anemia (41.6%), zinc deficiency (32.4%), and vitamin A deficiency (19.3%) all exceeded national averages and were highest in the 6-11 mo age category. The ENSANUT-ECU found high levels of nutrient intake inadequacies in the general population for protein, iron, and zinc. Rice comprises nearly one-third (32.8%) of energy in the diet, with relatively low levels of animal source foods. USFQ conducted the Chispaz Study examining the efficacy of a micronutrient powder; this study was carried out in Pastocalle. Thus, there is already an understanding and appreciation for research in the community.

Risks and Benefits. There are less than minimal risks associated with this study. The risk of an allergic reaction to eggs is low; expected to be only between 1 to 2% in young children. The majority of cases are mild consisting of hives soon after consuming eggs. Children with a known egg allergy will be excluded from the study and any children displaying any symptoms of an allergic reaction will be referred for treatment and will be excluded from any future participation in the study. There is a small risk associated with the blood draw for this study. The study team collecting samples will be well-trained on safe handling of human biologic specimens and will follow strict hygienic protocols relating to the usage of gloves, sterile equipment, and alcohol swabs to cleanse the area. A numbing cream is similarly being explored as an option to minimize pain for the child and psychological distress for the mother/caregiver. Interviews will be conducted with caregivers in a private setting to maintain confidentiality.

The children will benefit directly through their participation in this study through the likely improvements in nutritional status via consumption the consumption of eggs, a high nutritional quality, nutrient-dense food. The study involves a delayed intervention design, where eventually all participants will have the opportunity to receive the egg intervention. Thus, all participants have the opportunity to benefit through the receipt of a high quality food. There are potential benefits to society in terms of knowledge gained regarding a food-based, sustainable approach to improving young child nutrition. Globally, nutrition programming and policies have largely relied on the use of single nutrient or multiple nutrient supplementation, micronutrient powders, or imported processed complementary foods. This project aims to test a food-based approach, providing nutrients through eggs in a highly bioavailable matrix appropriate for young children. Further, the eggs are purchased locally with likely positive implications for economic development in the region.

Privacy and confidentiality. The consent, interview, anthropometric measurement, and blood draw processes will occur at community centers, health care posts or children nurseries -as the field team may determine the most appropriate location in each district of the parish. The spaces are sufficiently large to ensure confidentiality. Separate, private space in each of these settings will be designated for interviews and data collection. Only questions pertaining to child nutrition will be asked to avoid any unnecessary invasion of privacy. Additional time will be allocated for each consent and interview process to allow mothers/primary caregivers to ask additional questions as needed. They are also located in close proximity to households to facilitate convenient access for mothers and caregivers. In some cases, the field team will visit directly the participants at home for the purpose above mentioned.

The informed consent form will include mention of the possible use of data and blood samples for future research, as optional for consent on the part of mothers/caregivers. Two questions will be included in the baseline survey, the first asking if mothers/caregivers agree that their data may be used for future research and the second, asking mothers/caregivers if the blood of the child may be used for future research.

Data will be collected on paper forms and will be stored in locked cabinets in the Instituto de Investigacion en Salud y Nutricion (ISYN) office. All participants will be assigned a unique identifier that will be written on all study forms. Access to personal identifying information will be limited among the research investigators to only the PI, the senior research team, and the field team the purposes of participant follow-up and tracking. Data will be entered by the study team at USFQ. Encrypted raw data files will be transferred periodically to Washington University using password protected storage devices or other electronic data transfer mechanisms. De-identified datasets will be shared with co-PIs. In Ecuador, the study will be previously approved by the IRB (Comité de Bioética) of the USFQ and by the Ministry of Public Health.

ELIGIBILITY:
Inclusion Criteria:

* child is healthy and between the age of 6 months to 9 months

Exclusion Criteria:

* age of child
* any reactions to eating to eggs, a rash, hives, difficulty breathing

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Serum/plasma concentrations of B12, choline, and betaine | 6 months
  Venous blood collection
Serum/plasma concentrations of polyunsaturated fatty acids (PUFAs) and amino acids | 6 months
  Venous blood collection

SECONDARY OUTCOMES:
Attitudes, beliefs, and use of eggs in Pastocalle during the complementary feeding period. | 6 months
  Qualitative assessments: focus groups; in-depth interviews
Frequency of consumption of eggs, other animal source foods, and dietary diversity more broadly in the child's diet in Pastocalle. | 6 months
  Household survey

CONTACTS AND LOCATIONS:
Overall Officials: Lora Iannotti, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Pastocalle Parish, Pastocalle, Cotopaxi Province, Ecuador

REFERENCES:
- [Background] Charmaz, K, 1995, 'Grounded theory' in Rethinking methods in psychology.'
- [Background] Charmaz, K, 2000, 'Grounded theory: Objectivist and constructivist methods' in Handbook of qualitative research (2nd Edition).
- [Background] Charmaz, K, 2006, Constructing grounded theory: A practical guide through qualitative analysis.
- [Background] Clarke, A, 2005, 'Situational analysis: Grounded theory after the postmodern turn.'
- [Background] Davies, R, and Dart, J, 2005, The 'Most Significant Change' (MSC) Technique. Guide to Its Use Gibson RS. Principles of nutrition assessment. 2nd ed. New York: Oxford University Press; 2005.
- [Background] Guldan GS, Fan HC, Ma X, Ni ZZ, Xiang X, Tang MZ. Culturally appropriate nutrition education improves infant feeding and growth in rural Sichuan, China. J Nutr. 2000 May;130(5):1204-11. doi: 10.1093/jn/130.5.1204. PMID 10801920
- [Background] Hedeker D, Gibbons R. Longitudinal Data Analysis. 1st ed. Hoboken, NJ: Wiley, John & Sons, Incorporated; 2006.
- [Background] Iannotti LL, Lutter CK, Bunn DA, Stewart CP. Eggs: the uncracked potential for improving maternal and young child nutrition among the world's poor. Nutr Rev. 2014 Jun;72(6):355-68. doi: 10.1111/nure.12107. Epub 2014 May 7. PMID 24807641
- [Background] Jones KM, Ramirez-Zea M, Zuleta C, Allen LH. Prevalent vitamin B-12 deficiency in twelve-month-old Guatemalan infants is predicted by maternal B-12 deficiency and infant diet. J Nutr. 2007 May;137(5):1307-13. doi: 10.1093/jn/137.5.1307. PMID 17449597
- [Background] Lofland, J. and Lofland, L, 1995. Analyzing Social Settings: A Guide to Qualitative Observation and Analysis. Belmont, CA: Wadsworth.
- [Background] Institute of Medicine (US) Panel on Micronutrients. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222310/ PMID 25057538
- [Background] Pelto GH, Armar-Klemesu M, Siekmann J, Schofield D. The focused ethnographic study 'assessing the behavioral and local market environment for improving the diets of infants and young children 6 to 23 months old' and its use in three countries. Matern Child Nutr. 2013 Jan;9 Suppl 1(Suppl 1):35-46. doi: 10.1111/j.1740-8709.2012.00451.x. PMID 23167583
- [Background] Reichertz, Jo (2009). Abduction: The Logic of Discovery of Grounded Theory [39 paragraphs]. Forum Qualitative Sozialforschung / Forum: Qualitative Social Research, 11(1), Art. 13.
- [Background] Strauss and Corbin, 1994, 'Grounded theory methodology: An overview' in Handbook of qualitative research (1st Edition).
- [Background] Strauss and Corbin 1998, Basics of qualitative research: Grounded theory procedures and techniques (2nd Edition).
- [Background] Taneja S, Strand TA, Kumar T, Mahesh M, Mohan S, Manger MS, Refsum H, Yajnik CS, Bhandari N. Folic acid and vitamin B-12 supplementation and common infections in 6-30-mo-old children in India: a randomized placebo-controlled trial. Am J Clin Nutr. 2013 Sep;98(3):731-7. doi: 10.3945/ajcn.113.059592. Epub 2013 Jul 31. PMID 23902779
- [Background] World Health Organization (WHO). The WHO Child Growth Standards. Version current 1 April 2013. Internet: http://www.who.int/childgrowth/en/.
- [Background] World Health Organization (WHO). Indicators for assessing infant and young child feeding practices Part 1.
- [Derived] Evers EC, Waters WF, Gallegos-Riofrio CA, Lutter CK, Stewart CP, Iannotti LL. A sex- and gender-based analysis of factors associated with linear growth in infants in Ecuadorian Andes. Sci Rep. 2022 Feb 28;12(1):3292. doi: 10.1038/s41598-022-06806-3. PMID 35228574
- [Derived] Iannotti LL, Lutter CK, Waters WF, Gallegos Riofrio CA, Malo C, Reinhart G, Palacios A, Karp C, Chapnick M, Cox K, Aguirre S, Narvaez L, Lopez F, Sidhu R, Kell P, Jiang X, Fujiwara H, Ory DS, Young R, Stewart CP. Eggs early in complementary feeding increase choline pathway biomarkers and DHA: a randomized controlled trial in Ecuador. Am J Clin Nutr. 2017 Dec;106(6):1482-1489. doi: 10.3945/ajcn.117.160515. Epub 2017 Nov 1. PMID 29092879